CLINICAL TRIAL: NCT01558817
Title: Changing the Paradigm of In-Hospital Cardiopulmonary Resuscitation With Informed Assent: A Pilot Study
Brief Title: Changing the Paradigm of In-Hospital Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Renee Stapleton, Associatet Professor, Pulmonary and Critical Care Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PilotCPR001
Record Dates: First submitted 2012-02-21; First posted 2012-03-20 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-02

CONDITIONS: Oxygen Dependent COPD; Advanced Malignancy
Keywords: CPR; Palliative; Outcome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Informational brochure (Active Comparator): Patients receive an informational brochure
  Interventions: Behavioral: Informational Brochure
- Intervention (Experimental): Patients receive physician-directed informed assent intervention regarding CPR and informational brochure.
  Interventions: Behavioral: Informed Assent

INTERVENTIONS:
Behavioral: Informed Assent — Patients receive informed assent approach toward in-hospital CPR outcomes. Patients are informed that their underlying chronic illness makes outcomes after CPR so poor that CPR is not performed while allowing them to disagree.
  Arms: Intervention
Behavioral: Informational Brochure — An informational brochure about CPR will be given without a discussion with a physician.
  Arms: Informational brochure

SUMMARY:
Outcomes after in-hospital cardiopulmonary resuscitation (CPR) are very poor, particularly in patients with oxygen dependent chronic obstructive pulmonary disease (COPD) or metastatic cancer. Recent work found that in-hospital CPR is being performed more often before death with unchanging survival and that fewer CPR survivors are being discharged home, thus suggesting that CPR is increasingly performed without benefit and that the burden of this ineffective treatment is increasing. Unlike other medical procedures, CPR has become the default provided to all patients even those with tremendously poor outcomes. It is time to change the paradigm of CPR. Through comparing an innovative "informed assent" approach toward in-hospital CPR (informing patients that their underlying chronic illness makes outcomes of CPR so poor that CPR is not performed while allowing them to disagree) versus usual care in a group of chronically ill patients with reduced life expectancy, the investigators aspire to demonstrate that CPR delivery can be reduced. And in addition that DNR status increases, while preserving patient quality of life and decreasing the burden of this ineffective treatment to both patients and families. If effective, this informed assent intervention has the potential to revolutionize how the investigators discuss CPR with the investigators chronically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Oxygen dependent COPD or Advanced Malignancy
* Life expectancy of less than two years

Exclusion Criteria:

* Subjects who have already firmly decided to undergo CPR
* Subjects enrolled in a hospice program
* Subjects unable to speak English
* Subjects incapable of making their own decisions at the time of enrollment
* Subjects cared for by the study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Resuscitation Preference | Within couple of hours before the intervention and immediately (up to 2 days) after the intervention
  The primary outcome will be the difference in the proportion of patients in the informed assent intervention and informational brochure groups reporting preferences to be DNR (do not rescusitate).

SECONDARY OUTCOMES:
Depression | Baseline (day of intervention) and 2 weeks after intervention
  Patients' and family members' symptomes of depression will be measured by the PHQ-8 questionnaire.
Anxiety | Baseline (day of intervention) and two weeks after intervention
  Patients and families will complete the GAD-7 questionnaire, a measure of generalized anxiety disorder.
Physician Order for Life Sustaining Treatment (POLST) | Baseline (day of intervention) and 2 weeks after intervention
  Participants who expressed a preference to be DNR will be asked to complete a POLST form by their physician. It will also be explained that this can be changed any time the status changes.
DNR status preference | Two weeks after the intervention
  The difference in DNR status preference between patients in the control and invervention group at two weeks after the intervention.
Report on acceptability of the informed assent approach | Within couple of hours (up to 2 weeks) after intervention
  The following questions will be asked:
  1. How helpful was this approach to discussing CPR with respect to CPR decisions?
  2. Would you recommend this approach to discussing CPR for other patients who have serious illnesses?
Assessment of DNR status change or intervention follow-up from primary physician | Three months after the intervention
  Contact the physician for each patient at 3 months after the study visit to determine whether there are changes in the DNR status or if the physician has talked with the patients about the status since the study visit.
Resource utilization | Up to 6 months after intervention or until death
  Record resource utilization for participants that includes hospitalizations, ICU care, use of hospice etc by medical record review.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Vermont and Fletcher Allen Health Care, Burlington, Vermont
  - University of Washington, Seattle, Washington